CLINICAL TRIAL: NCT04852796
Title: Efficacy and Safety of the Anti- COVID-19 Vaccin in Clinical Hematology Patients
Acronym: HEMVACO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cornouaille (Other)
Responsible Party: Sponsor
Other Study IDs: QP2021-PPD
Record Dates: First submitted 2021-03-30; First posted 2021-04-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Covid19; Hematologic Malignancy; Vaccine Response Impaired
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with hemopathy — optimal humoral response at 1 month after COVID-19 vaccination

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an emerging infectious disease that was first reported in December 2019 in Wuhan, China. Infection with this new coronavirus called SARS-CoV-2 can lead to fatal pneumonia associated with high rates of hospitalization in intensive care units (ICU).

Hospitalized patients with hematologic malignancies have a higher mortality rate than patients without hematologic malignancies (62% vs. 8%). The severity of Covid-19 may be related to their treatment, in particular anti-CD20 used in B lymphoid hemopathies. In fact, anti-CD20 antibodies induce rapid and prolonged depletion of B cells, but they are necessary for development. humoral immune responses.

But currently, no immunogenicity data are known for patients with hemopathy or in those on anti-lymphocyte immunochemotherapy.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the humoral response after vaccination against SARS-CoV-2 in a French multicenter cohort of patients with hemopathies. Analysis of hemopathies and immunochemotherapy subgroups will determine whether there is a need to strengthen immunization schedules. In addition, the study wish to assess the safety and clinical efficacy of mRNA vaccines in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Benign or malignant hemopathy
* With priority vaccination indication
* Having benefited from anti-covid-19 mRNA vaccination

Exclusion Criteria:

* Patients under legal protection
* Palliative care patients
* History of known Covid-19 disease (<1 year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemopathy followed in declared hospitals
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
humoral response after COVID19 vaccination | 1 month after vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)

SECONDARY OUTCOMES:
humoral response after COVID19 vaccination | before first dose vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)
humoral response after COVID19 vaccination | before second dose vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)
humoral response after COVID19 vaccination | 3 months after vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)
humoral response after COVID19 vaccination | 6 months after vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)
humoral response after COVID19 vaccination | 12 months after vaccination
  SARS-CoV-2 Trimeric S IgG titers (BAU/ml)
clinical response after COVID19 vaccination | 12 months after vaccination
  SARS-CoV-2 disease onset in the follow-up
security of mRNA COVID19 vaccine | 3 months after vaccination
  side effects onset in the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: LENAIG LE CLECH, PhD, Principal Investigator — Centre Hospitalier de Quimper Cornouaille
Locations (1):
- Centre Hospitalier de Quimper Cornouaille, Quimper, France

REFERENCES:
- [Derived] Gueguen M, Khatchatourian L, Loheac C, Dorval I, Mercier M, Le Calloch R, Mahe K, Rizcallah MJ, Hutin P, Fangous MS, Saidani N, Le Clech L. The humoral response of mRNA COVID-19 vaccine in hematological diseases: The HEMVACO study. Infect Dis Now. 2022 Aug;52(5):280-285. doi: 10.1016/j.idnow.2022.05.008. Epub 2022 Jun 3. PMID 35667558